CLINICAL TRIAL: NCT02211248
Title: Cardiovascular Autonomic Control Evaluation Through Cardiac Frequency Variability in Hypertensive Patients Subjected to Distinct Interventions: Clinical Trial
Brief Title: Cardiovascular Autonomic Control Evaluation Through Cardiac Frequency Variability in Hypertensive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Silvia Goldmeier, Doctor, Instituto de Cardiologia do Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4524/10
Record Dates: First submitted 2014-07-31; First posted 2014-08-07 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Hypertension
Keywords: Cardiac Frequency Variability; multidisciplinary care; clinical trial
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional Group (Active Comparator): Conventional treatment and follow up
  Interventions: Other: Conventional treatment and follow up
- Multidisciplinary Group (Experimental): Multidisciplinary assistance
  Interventions: Other: Multidisciplinary assistance

INTERVENTIONS:
Other: Multidisciplinary assistance — Multidisciplinary group assistance was effected every two months by all professionals (physician, nurse, dietitian, physiotherapist and psychologist) and consisted in orientations and mechanisms to medication and non-pharmacological adherence (lifestyle changes).
  Arms: Multidisciplinary Group
Other: Conventional treatment and follow up — Assistance was effected by physician and nurse and consisted about adapting to the drug
  Arms: Conventional Group

SUMMARY:
Analyzing cardiovascular evaluation measures in the multidisciplinary and in the conventional treatment of hypertensive patients will provide better parameters for comparing the two approaches.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years of age
* Diagnosis of primary hypertension

Exclusion Criteria:

* Neurological condition
* Cardiac condition
* Renal condition
* Congenital conditions
* Previous myocardial revascularization surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-12; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Cardiac Frequency Variability at 1 year | Measured at the first appointment and 1 year later

SECONDARY OUTCOMES:
Change from Baseline in Systolic and Diastolic Blood pressure | Measured at the first appointment and 1 year later

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Cardiologia do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil